CLINICAL TRIAL: NCT03338751
Title: Determine the Effect on Cognitive Impairment Measures by Providing Hearing-Assistance to Skilled Nursing Facility Residents
Acronym: DECIPHER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unfunded Pilot Study
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-00697
Record Dates: First submitted 2017-10-27; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Hearing Impairment
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hearing Assistance Device (HAD) First (Active Comparator): Tablet, loaded with REDCap will generate a random number that determines the order of test administration with the HAD first or second. Participants randomized to HAD first will use a Hearing Aid Device.
  Interventions: Diagnostic Test: cognitive testing with HAD (PockeTalker) First; Diagnostic Test: Cognitive testing without HAD First
- No Hearing Assistance Device (HAD) First (Active Comparator): Sham hearing aid device
  Interventions: Diagnostic Test: cognitive testing with HAD (PockeTalker) First; Diagnostic Test: Cognitive testing without HAD First

INTERVENTIONS:
Diagnostic Test: cognitive testing with HAD (PockeTalker) First — tablet, loaded with REDCap will generate a random number that determines the order of test administration with the HAD first or second.
  Other Names: PockeTalker Hearing Aid Device
Diagnostic Test: Cognitive testing without HAD First — tablet, loaded with REDCap will generate a random number that determines the order of test administration with the HAD first or second.

SUMMARY:
The purpose of the study is to see if a commercially available hearing assistance device called the PockeTalker has an effect on performance on cognitive (memory and thinking) tests among skilled nursing facility residents.

Investigators are asking residents to perform cognitive tests with and without hearing assistance equipment known as PockeTalkers. This study will be conducted at one urban Skilled Nursing Facility (SNF) with the goal of understanding the extent to which hearing impairment impacts commonly used cognitive impairment measures for clinical assessment. Cognitive performance will be measured, cerumen occlusion, and perceived hearing.

ELIGIBILITY:
Inclusion Criteria:

* admitted to unit of intervention
* ability to communicate and follow simple commands
* capacity to consent assessed with standard questions used to assess capacity or having a surrogate who can provide consent.

Exclusion Criteria:

* not on the unit of intervention
* obtunded or comatose state
* inability to communicate verbally
* inability to consent and without surrogate
* non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Measure of Cognitive function using Mini-Cog | 20 Minutes
  three-item recall and a clock draw test. 24 Medical assistants have been trained and have employed this test successfully in primary care practices. The Mini-Cog has test characteristics that are comparable to any other brief instrument and exceeds most in accuracy or predictive quality.
Perceived Hearing measured by Hearing Handicap Inventory for the Elderly-Screening Version (HHIE) | 20 Minutes
  HHIE-S is a valid, robust test for identifying hearing-impaired elderly, irrespective of the audiometric definition used to finally diagnose hearing difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Chodosh, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided